CLINICAL TRIAL: NCT07371117
Title: Effect Of Silverdiamine Fluoride Gel, Sodium Fluoride With CPP-ACP, APF On Early Childhood Caries - A Randomised Controlled Trial
Acronym: SDF
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Renuga Lakshmi Apathsakayan, Assistant Professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CODJU-21041
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Early Childhood Caries (ECC); Dental Caries
Keywords: silver diamine fluoride
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride; Sodium Fluoride; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Intervention Model Description: This three-arm phase 2 clinical trial will be conducted to evaluate the effectiveness of silver diamine fluoride (SDF) for preventing or arresting dental caries.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cavitated/Non cavitated caries lesions involving only enamel (Experimental): Reversible pulpitis
  Interventions: Drug: Silver Diamine Fluoride (SDF, 38%); Drug: Sodium Fluoride with CPP-ACP; Drug: Acidulated phospahate fluoride gel 1.23%
- Experimental arm including cavitated/ non cavitated caries lesions involving enamel,dentin but not p (Active Comparator)
  Interventions: Drug: Silver Diamine Fluoride (SDF, 38%); Drug: Sodium Fluoride with CPP-ACP; Drug: Acidulated phospahate fluoride gel 1.23%

INTERVENTIONS:
Drug: Silver Diamine Fluoride (SDF, 38%) — Silver diamine fluoride gel is applied in gel form
Drug: Sodium Fluoride with CPP-ACP — This is in a Topical fluoride varnish
Drug: Acidulated phospahate fluoride gel 1.23% — This is a topical fluoride application for 1 minute application

SUMMARY:
Early Childhood Caries (ECC) remains a global public health concern, necessitating minimally invasive, fluoride-based alternatives to conventional restorative therapy. Silver Diamine Fluoride (SDF), Sodium Fluoride with Casein Phosphopeptide-Amorphous Calcium Phosphate (NaF + CPP-ACP), and Acidulated Phosphate Fluoride (APF) gel are widely employed chemotherapeutic agents; however, comparative clinical evidence of their effectiveness in ECC management remains limited.

This randomized controlled clinical trial will evaluate and compare the efficacy of SDF gel, NaF + CPP-ACP, and APF gel in arresting and preventing ECC.

ELIGIBILITY:
Inclusion Criteria:

* The participants who had at least one untreated cavitated active caries lesion with dentin exposed based on the Nyvad criteria (level 3: "Enamel/dentin cavity easily visible with the naked eye where the surface of cavity feels soft or leathery on gentle probing", characterized by dentin exposure without signs of pulp involvement, pain, abscess, sinus tract, or mobility.
* Medically healthy children with no systemic disorders or developmental anomalies

Exclusion Criteria:

* Parents refused consent for study
* Any child with special health care needs or with any systemic ailments will be excluded from the study
* Teeth exhibiting irreversible pulpitis, abscess, pathological mobility, pathological radiographic changes

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dental caries arrest | Caries arrest will be assessed 6 months after intervention
  A lesion was considered active if a blunt dental probe penetrated the dentinal surface easily, whereas arrested caries resisted probe penetration, indicating surface hardening.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, jazan University, Jizan, Jazan Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the IPD because we consider to continue the study for long term in future